CLINICAL TRIAL: NCT01103440
Title: A Randomized, Pilot, Single-center Study, Investigator-Initiated Study to Look at an Aggressive Therapeutic Approach in Aspirin Resistant Patients Comparing to Standard for Patient Undergoing Percutaneous Coronary Intervention
Brief Title: Aspirin Resistance and Percutaneous Coronary Intervention (PCI)
Acronym: RESIST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Annapoorna Kini, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO-07-0200
Record Dates: First submitted 2010-04-12; First posted 2010-04-14 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-01

CONDITIONS: Stable Angina
Keywords: Major Adverse Cardiovascular Event; MACE; Death; MI; CK MB greater 3x Normal; Urgent Revascularization; Stent Thrombosis; Bleeding
MeSH Terms: conditions — Angina, Stable; Death; Hemorrhage | interventions — Clopidogrel; cangrelor; Abciximab; Eptifibatide; Tirofiban; Thienopyridines; Ticlopidine; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Conventional Strategy (Other): Patient receive 325 mg ASA orally and loading does of 600mg Clopidogrel at time of procedure
  Interventions: Drug: Antiplatelet Therapy (ASA, Clopidogrel)
- Aggressive Strategy (Active Comparator): Patient receive 325mg ASA orally and loading does of 600mg Clopidogrel at time of procedure with addition of IV GP IIb/IIIa inhibitor bolus intra procedurally
  Interventions: Drug: Intravenous Glycoprotein inhibitor + ASA, Clopidogrel

INTERVENTIONS:
Drug: Intravenous Glycoprotein inhibitor + ASA, Clopidogrel — IV Glycoprotein IIb/IIIa inhibitor bolus intra procedurally
  Other Names: Cangrelor; Abciximab; Eptifibatide; Tirofiban
  Arms: Aggressive Strategy
Drug: Antiplatelet Therapy (ASA, Clopidogrel) — Standard antiplatelet PCI treatment
  Other Names: Thienopyridines; Ticlopidine; Clopidogrel; Prasugrel
  Arms: Conventional Strategy

SUMMARY:
The objective of this study is to evaluate if aggressive antiplatelet therapy would reduce ischemic events in aspirin (ASA) resistant patients after percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
This is the first US based randomized double blinded prospective study using triple antiplatelet therapy and double dose plavix maintenance dose in aspirin resistant patients undergoing elective PCI through femoral access. The primary outcome of this study is an elevation of cardiac enzymes within 24 hours after the PCI with a secondary outcome of a composite of major adverse cardiac events of death, MI, stent thrombosis and urgent revascularization and bleeding up to 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* Scheduled for elective or ad-hos PCI
* Aspirin use daily for greater or equal to one week
* Aspirin resistant (ARU greater than or equal to 550 on Verify Now-ASA

Exclusion Criteria:

* Pre-procedural elevation of cardiac biomarkers (CK-MB greater or equal to 10.4ng/dl or Tnl greater or equal to 0.4ng/dl
* administration of any GP IIb/IIIa inhibitor, anticoagulation or lytic therapy in the previous 30 days
* Ongoing bleeding or bleeding diathesis, contraindications for anticoagulation or increased bleeding risk or history of bleeding in the last eight weeks
* Previous stroke or transient ischemic attack or any intracranial pathology in the last six months, major surgery or trauma within the previous six weeks
* Platelet count less than hundred thousand per cubic millimeter or hematocrit <33% or hemoglobin <11 g per deciliter
* Subjects who received full dose low molecular weight heparin within six hours prior to randomization
* Allergy or intolerance to any of the study drugs or the presence of any serious comorbidity with life expectancy of ≤1year
* Scheduled for saphenous vein graft intervention, chronic total occlusions or with impaired renal function (eGFR<60ml/min) or patients who were taking anticoagulants or antiplatelet agents other than aspirin and clopidogrel or nonsteroidal anti-inflammatory drugs within two weeks before the PCI procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annapoorna S Kini, MD MRCP, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 330 patients were screened with 36 enrolled between April 2007 and December 2008
Period: Overall Study
Arm/Group | Conventional Strategy | Aggressive Strategy
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Strategy | Aggressive Strategy | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (10) | 66.2 (9) | 65.7 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Elevation of Cardiac Enzyme
Description: Number of participants with peri-procedural biomarker elevation defined as any elevation above baseline of CK-MB or Tn-I within 24 hours after completion of the procedure.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Strategy | Aggressive Strategy
Number analyzed (Participants) | 18 | 18
Participants | 4 | 2

2. Secondary Outcome: Number of Participants With Major Adverse Cardiac Event (MACE)
Description: Number of participants with MACE which is any event of Death, MI, Stent Thrombosis, Urgent Revascularization, Bleeding. Major adverse cardiac events (MACE), defined as the composite of death, MI (CK-MB > 3 times normal), urgent revascularization and definite or probable stent thrombosis (ST) within 30 days. Stent thrombosis was defined according to the new academic research consortium definitions; 2) bleeding complications within 30 days. Major bleeding was defined as intracranial or intraocular bleeding or a drop in hemoglobin > 5 g/dL. Minor bleeding was defined as hemorrhage at the access site requiring intervention, hematoma with a diameter of at least 5 cm, a reduction in hemoglobin levels of at least 4 g/dL without an overt bleeding source or at least 3 g/dL with such a source, reoperation for bleeding or transfusion of a blood product.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Strategy | Aggressive Strategy
Number analyzed (Participants) | 18 | 18
Participants | 5 | 1

ADVERSE EVENTS:
Arm/Group | Conventional Strategy | Aggressive Strategy
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 15/18 | 4/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conventional Strategy (N=18) | Aggressive Strategy (N=18)
Stent thrombosis (Cardiac disorders) | 2 | 0
Urgent Vascularization (Cardiac disorders) | 2 | 0
Myocardial Infarction (Cardiac disorders) | 2 | 0
Major Bleeding (Blood and lymphatic system disorders) | 1 | 0
Minor Bleeding (Blood and lymphatic system disorders) | 2 | 1
Cardiac Enzyme Elevation: Troponin-I (Cardiac disorders) | 4 | 2
Cardiac Enzyme Elevation: CK-MB (Cardiac disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
Small pilot study with a limited sample size and not powered to detect differences in individual ischemic endpoints. Study does not delineate an optimal dose of aspirin. Antiplatelet effect of aspirin may fluctuate in patients at the same dosage.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes